CLINICAL TRIAL: NCT05673655
Title: Evaluation of Ultrasound Sonography Intraoral Guided Injection of Botulinum Toxin in Masseter Muscle
Brief Title: Intraoral Injection of Trigger Points by Botox
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohsen, principal investigator, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC2213
Record Dates: First submitted 2023-01-04; First posted 2023-01-06 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Myofacial Pain
MeSH Terms: conditions — Facial Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transcutaneous injection (Active Comparator)
  Interventions: Drug: transcutaneous trigger point injection by botox
- intraoral injection (Active Comparator)
  Interventions: Drug: intraoral trigger point injection by botox

INTERVENTIONS:
Drug: intraoral trigger point injection by botox — intraoral injection of trigger point of masseter muscle by botulinum toxin
  Arms: intraoral injection
Drug: transcutaneous trigger point injection by botox — transcutaneous injection of masseter muscle by botulinum toxin
  Arms: transcutaneous injection

SUMMARY:
Patients with orofacial pain lasting at least 3 months. The patients will be randomly assigned to one of the two groups according to the treatment method: group I (intraoral injection) and group II (transcutaneous injection) where each patient injected Botox at each trigger point according to the treatment group by the same operator. Patients will be examined by a blinded investigator at pre- and post-injections at the following intervals: during diagnosis, 1 week, 4, and 6 weeks post-injection. The patients will be assessed using a pain score measured on a 10-point visual analog scale (VAS). The secondary outcome assessed will be measuring the quality of life in an Oral Health Impact Profile questionnaire (OHIP-14).

ELIGIBILITY:
Inclusion Criteria:

* Definite diagnosis of myofascial pain with a referral
* the presence of one or more trigger points in the unilateral or bilateral masseter muscle -
* no history of any invasive procedures in the related masseter muscle

Exclusion Criteria:

* Factors that can cause pain in the orofacial region other than trigger points (decayed tooth, temporomandibular joint internal disorder).
* Any systemic disease that possibly affects the masticatory system such as rheumatoid arthritis and epilepsy
* pregnancy and lactation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-25 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-02-25 (Estimated)

PRIMARY OUTCOMES:
pain score | 6 weeks post injection
  The participated patients will be assessed using pain score measured on a 10-point visual analogue scale (VAS), the 0 indicating no pain and 10 indicating the worst pain ever.

SECONDARY OUTCOMES:
(OHIP-14) scale | 6 weeks
  OHIP-14 is used to measure patients' self-reported discomfort, disability, and functional limitation due to oral conditions with scores ranging from 0 to 56 (with 56 representing a subject answering ''very often'' to all 14 items

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University, Al Fayyum, Egypt

REFERENCES:
- [Derived] Shabaan AA, Kassem I, Aboulmagd I, Amer IA, Shaaban A, Abd-El-Ghafour M, Refahee SM. Effectiveness of intra-oral botulinum toxin injection in comparison to the extra-oral approach on pain and quality of life in patients with myofascial pain: a randomized clinical trial. Clin Oral Investig. 2024 Dec 17;29(1):18. doi: 10.1007/s00784-024-06051-0. PMID 39681752